CLINICAL TRIAL: NCT05271292
Title: A Phase 1b/2, Single-Arm, Open-Label, Dose-Escalation, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Chiauranib for the Treatment of Advanced Solid Tumors and Relapsed/Refractory SCLC
Brief Title: Chiauranib for Advanced Solid Malignant Tumors and Relapsed/Refractory SCLC.
Acronym: SCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAR107
Record Dates: First submitted 2022-01-26; First posted 2022-03-09 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Small Cell Lung Cancer; Advanced Solid Malignant Tumor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — chiauranib

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled sequentially in 3 dose-escalating cohorts (Chiauranib capsules 35mg, 50 mg and 65 mg once daily)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study arm (35 mg) (Experimental): Phase 1b: Patients will be enrolled sequentially in 3 dose-escalating cohorts (Chiauranib capsules 35, 50, and 65 mg, orally)
  Interventions: Drug: Chiauranib
- Study arm (50 mg) (Experimental): Phase 1b: Patients will be enrolled sequentially in 3 dose-escalating cohorts (Chiauranib capsules 35, 50, and 65 mg, orally)
  Interventions: Drug: Chiauranib
- Study arm (65 mg) (Experimental): Phase 1b: Patients will be enrolled sequentially in 3 dose-escalating cohorts (Chiauranib capsules 35, 50, and 65 mg, orally)
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — Phase 1b: Each patient will undergo both a single-dose period (6 days) and a consecutive-dose (1 cycle of 28 days) period
  Phase 2: Patients will take the RP2D once daily for 28-day cycles continuously with no interruption between cycles
  Other Names: CS2164

SUMMARY:
This is a Phase 1b/2, single-arm, open-label, dose-escalation study including 2 stages:

Phase 1b: Dose-Escalation Stage (Single-Dose and Consecutive-Dose Periods)

Phase 2: recommended Phase 2 dose (RP2D) of chiauranib will be given to all patients enrolled in this phase once daily for 28-day cycles continuously with no interruption between cycles.

DETAILED DESCRIPTION:
Phase 1b:

Patients with advanced solid malignant tumor (including SCLC, NSCLC, colorectal carcinoma, pancreatic carcinoma, hepatocellular carcinoma, ovarian cancer, neuroendocrine tumors, non-Hodgkin's lymphoma and others) that has relapsed from or is refractory to standard therapy or for which no standard therapy exists will be enrolled to the 35 mg, 50 mg and 65 mg dose cohorts in this stage. The starting dose is 35 mg, and each higher dose cohort will not enroll until the lower dose is deemed safe.

After screening, eligible patients will be enrolled sequentially in 3 dose-escalating cohorts. Based on an estimated average body weight of 60 kg, the initial dose of chiauranib will be 35 mg once daily, and the dose will be escalated to 50 mg and 65 mg once daily, depending on the occurrence and frequency of DLTs. The 3+3 design will be employed in dose escalation decisions.

Each dose cohort will enroll at least 3 patients. Overenrolling dosing cohorts is allowed to allow for potential screen failures and/or subjects who end up being not evaluable by not completing the DLT evaluation period. Each subject will undergo both a single-dose period (6 days) and a consecutive-dose (1 cycle of 28 days) period, as described below. DLTs will be evaluated during this period (a total of 34 days).

Phase 2:

SCLC patients with progressive disease or recurrence after at least 2 previous regimens, including one platinum-based chemotherapy, will be enrolled in this stage. The RP2D will be given to all subjects enrolled in this stage. Subjects will take the RP2D chiauranib once daily for 28-day cycles continuously with no interruption between cycles.

ELIGIBILITY:
Phase 1b

Inclusion Criteria:

1. Patient is at least 18 years of age, regardless of gender. Patient has a diagnosis of histologically or cytologically confirmed advanced solid malignant tumor (including SCLC, NSCLC, colorectal carcinoma, pancreatic carcinoma, hepatocellular carcinoma, ovarian cancer, neuroendocrine tumors, non-Hodgkin's lymphoma, and others) that has relapsed from or is refractory to standard therapy or for which no standard therapy exists.
2. Patient has at least one measurable target lesion as defined by RECIST1.1, i.e., a lesion that has radiologic evidence of disease progression, after treatment with radiotherapy or local-regional therapy.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 at enrollment.
4. Major organ functions meet the following criteria (no corrective treatment, such as G CSF, erythropoietin, and blood transfusion, within 2 weeks before enrollment):

   1. Hematology: absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥100 g/L.
   2. Biochemistry: total bilirubin ≤1.25×upper limit of normal (ULN), both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN (≤5×ULN for patients with hepatic metastasis), creatinine clearance >60 mL/min (according to Cockcroft-Gault equation), fasting triglyceride ≤3.0 mmol/L, fasting total cholesterol ≤7.75 mmol/L.
   3. Coagulation panel: international normalized ratio (INR) <1.5.
5. Patient has a life expectancy ≥3 months.
6. Patient is able to provide voluntary informed consent.
7. Women of childbearing potential (WOCBP) must be willing and able to take highly effective contraceptive measures during the entire study treatment period and for 12 weeks after the last dose of study drug (see Appendix 11.7). Women of childbearing potential include premenopausal and not sterilized (by hysterectomy, bilateral ligation of fallopian tubes, or bilateral oophorectomy) females who have passed menarche.
8. Male patients must be willing and able to use male condoms and their female partners who are WOCBP during the entire study treatment and for the 12 weeks after the last dose of the study drug.

Exclusion Criteria:

1. Patient has received any systemic anticancer therapy (including chemotherapy, targeted therapy, biological immunotherapy, any investigational drug, or anti-cancer herbal medicine) within 21 days before enrollment, or any blood support therapy (including blood transfusion, blood products, or hematopoiesis stimulating agents such as granulocyte-colony stimulating factor [G-CSF]) within 2 weeks before enrollment.

   a. Patients who are receiving corticosteroids at a dose of > 10 mg prednisone or equivalent of other systemic steroids will be excluded.
2. Patient with prior or concurrent malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of investigational regimen.
3. Patient has uncontrolled or significant cardiovascular diseases, including:

   1. New York Heart Association (NYHA) grade II or higher congestive cardiac failure, unstable angina pectoris, and/or myocardial infarction within the 6 months prior to the first dose of the investigational drug, clinically significant arrhythmia unable to be controlled with medical treatment or left ventricular ejection fraction (LVEF) < 50% at screening.
   2. Primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy).
   3. Clinically significant history of prolonged QTc interval, or QTcF interval >470ms for females or >450 ms for males during screening.
   4. Coronary heart disease with symptoms requiring medication.
4. Patient has hypertension at screening (defined as systolic blood pressure [SBP] ≥140 mmHg, diastolic blood pressure [DBP] ≥90 mmHg). (Patients with a known history of hypertension if blood pressure is considered well controlled on a single anti-hypertensive medication (systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg at screening) and in whom there has been no change in blood pressure medication for 3 months prior to screening due to poor control.)
5. Patient has active hemoptysis, has had active bleeding within 6 months prior to enrollment, or has definite predisposition to gastrointestinal bleeding as determined by the investigator (e.g., esophageal varix associated with bleeding risk, local active ulcer lesions).
6. Patient has uncontrolled pleural effusion, hydropericardium, or ascites.
7. Patient has active or symptomatic central nervous system (CNS) metastases that require treatment.
8. Patient has a history of deep vein thrombosis, pulmonary embolism, or other serious thrombotic event within 6 months prior to enrollment.
9. Patient has an interstitial lung disease (ILD) that requires treatment, such as idiopathic interstitial pneumonia, pulmonary fibrosis, or evidence of ILD in baseline chest computed tomography (CT) or magnetic resonance imaging (MRI).
10. Patient has any current toxicity (except alopecia) of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, Grade 2 or higher caused by previous therapy.
11. Patient has clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of the study drug (e.g., inability to swallow, chronic diarrhea, intestinal obstruction), or has had total gastrectomy, according to the investigator's judgment.
12. Patients has undergone a major surgical operation within 6 weeks prior to screening or a minor surgical operation within 2 weeks prior to screening. A major surgical operation refers to an operation involving general anesthesia but excludes procedures such as endoscopies for diagnostic purpose or an implantation of vascular access devices.
13. Patient has urine protein ≥2+ by urine routine examination and urine protein ≥1 g/24 h by 24-hour urine protein quantification.
14. Patient has serious active infection or known infectious disease including hepatitis B, hepatitis C infection in active stage, or HIV/AIDS.
15. Patient has any mental or cognitive impairment that may limit their understanding and implementation of written informed consent and compliance in this study.
16. Patient has previously experienced toxicity leading to discontinuation of treatment with Aurora kinase inhibitors or VEGF/VEGFR inhibitors, such as sorafenib, sunitinib, pazopanib, bevacizumab, regorafenib, axitinib, vandetanib, or dasatinib.
17. Patient has current drug or alcohol abuse disorders that may affect study participation, according to the investigator's judgment.
18. Women who are pregnant, planning to become pregnant, lactating, or who have positive pregnancy test results at screening or before the first dose.
19. Patients who are currently taking and have to continue taking strong CYP3A4 inhibitor drugs, such as ketoconazole, itraconazole, clarithromycin, telithromycin, nefazodone, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, or tipranavir, as well as strong CYP3A4 inducers, such as rifampin, dexamethasone, carbamazepine, during Phase 1b (dose escalation stage) of the study.
20. Any other conditions that make the patient inappropriate for participation in this study, at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and other safety parameters | Until 30 days after a patient takes the last dose of the study drug
  Number of patients experienced AEs
Incidence and characteristics of DLTs | 34 days
  Number of patients experienced any dose limited toxicity
MTD and recommended Phase 2 dose (RP2D) | 34 days
  Determination of recommended phase II dose

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Maximum plasma concentration (Cmax) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Area under the plasma concentration-time curve from 0 to infinity (AUC 0-inf) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Half-life (t½) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Trough plasma concentration (Cmin) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Area under the plasma concentration-time curve (AUC0-t) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Oral clearance (CL/F) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
accumulation ratio | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Steady state plasma concentration (Css) | Phase 1b: days 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles. Phase 2: days 1, 14, 28 during Cycle 1; and day 28 in Cycle 2 and all subsequent cycles (all cycles in phase 1b and 2 are 28 days each)
  PK Profile
Objective response rate (ORR) | 6 months
  preliminary efficacy of chiauranib
disease control rate (DCR) | 6 months
  preliminary efficacy of chiauranib
duration of response (DoR) | 6 months
  preliminary efficacy of chiauranib
progression-free survival (PFS) | 6 months
  preliminary efficacy of chiauranib
overall survival (OS) | 6 months
  preliminary efficacy of chiauranib
Correlation between ATRX gene mutation and efficacy | 6 months
  Efficacy outcomes in patients with ATRX gene mutation and wild-type respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Cabilia Pichardo, MD, Study Director — Executive Director of Clinical Development
Locations (11):
- United States (11):
  - California Cancer Associates-Encintas, Encinitas, California
  - Providence/St. Joe Cancer Institute/Crosson Cancer Institute, Fullerton, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institue, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Gabrail Cancer Center Research, Canton, Ohio
  - OU Health, Oklahoma City, Oklahoma
  - Sarah Cannon Research Center, Nashville, Tennessee
  - North Houston Cancer Clinics, Huntsville, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Meerbeeck JP, Fennell DA, De Ruysscher DK. Small-cell lung cancer. Lancet. 2011 Nov 12;378(9804):1741-55. doi: 10.1016/S0140-6736(11)60165-7. Epub 2011 May 10. PMID 21565397